CLINICAL TRIAL: NCT05388110
Title: Neurobiological Mechanism of SKY Breath Intervention
Brief Title: SKY Breath Intervention
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 21-33230
Record Dates: First submitted 2022-04-22; First posted 2022-05-24 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Depression; Anxiety Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Passive drool/saliva will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls
  Interventions: Behavioral: SKY Breath Intervention
- Depressed adolescents
  Interventions: Behavioral: SKY Breath Intervention

INTERVENTIONS:
Behavioral: SKY Breath Intervention — Sudarshan Kriya Yoga (SKY) is a breath-based meditative practice that entails a sequence of specific breathing techniques to help practitioners achieve a state of calm alertness. It has offered benefits as a therapeutic option for mild-to-moderate depression and anxiety disorders and as an adjunctive treatment in patients with major depressive disorder, but the neurological mechanism of SKY breath intervention is still not fully understood.

SUMMARY:
Depression is highly debilitating and prevalent among adolescents. Adolescent-onset depression is associated with long, severe, and recurrent episodes that are often not responsive to treatment. There is a dire need to develop novel treatments that are efficient, cost-effective, and tolerant for this population. Sudarshan Kriya Yoga (SKY) is a breath-based meditative practice that entails a sequence of specific breathing techniques to help practitioners achieve a state of calm alertness. It has offered benefits as a therapeutic option for mild-to-moderate depression and anxiety disorders and as an adjunctive treatment in patients with major depressive disorder, but the neurological mechanism of SKY breath intervention is still not fully understood.

The goal of this study is to determine the efficacy of SKY breath intervention in treating depressed adolescents and to understand its mechanisms. In this study, thirty depressed adolescents and thirty healthy controls will be recruited to evaluate the efficacy of the 8-week SKY intervention. Assessment for depression and anxiety, salivary cortisol, resting heart rate, blood pressure, and neuroimaging will be collected at the baseline, 4 weeks into SKY intervention (questionnaires only), and post-intervention.

This will be the first study to evaluate the potential benefits of of SKY breath intervention as a treatment option for depressed adolescents.

DETAILED DESCRIPTION:
Participants & Screening: All participants (16-24yrs) will be first screened for COVID and only those who are negative will be allowed to enroll. Participants who meet the criteria for the study at initial online screening will complete measures with study investigator including relevant demographics information and the BDI-II.

SKY Intervention: The SKY breath intervention will take place online via Zoom over 6 consecutive days for 3 hours each day as part of the Campus SKY Breath Meditation workshop.

Weekly intervention follow-ups: After completion of the 6-day online workshop, participants will be encouraged to continue a home-based practice (25 minutes per day, daily records is needed for reimbursement) and required to attend 1-hour weekly (online) follow-ups for 8 weeks during which there will be group practice of the workshop material. Attendance is mandatory for all follow-ups. Given the popularity of the program, participation is typically high. Instructor will verify attendance and ensure that all participants are proficient in performing SKY. The effectiveness of SKY and staying on track with study procedures are facilitated by subjects, therefore, the study consent will ask subjects if they are willing to share their email/phone with others in the study.

Cortisol Levels and Resting Heart Rate: During each MRI visit, saliva cortisol, blood pressure, and resting heart rate will be measured in participants. Passive drool/ saliva will be collected. Following this, subjects will do belly breathing exercise for 3-5 mins. Subjects will sit in a chair, and place one hand on the upper chest and the other hand on the belly. Subjects will be asked to breathe in slowly through the nose so they can feel their stomach rise, then will be asked to exhale slowly through their pursed lips so they can feel the hand on their chest remain relatively still. Saliva will then be collected in a microcentrifuge tube for 2 min and stored in a -80°C freezer in order to assess salivary cortisol levels. For measurement of cortisol, saliva will be assayed using a High-Sensitivity Salivary Cortisol Enzyme Immunoassay Kit from Salimetrics, Inc. Samples will be processed in a standard Bio-safety level 2 laboratory equipped to handle clinical samples with all the appropriate personal protective equipment. Not only is saliva collection less invasive than blood but it is also a routinely established method to assess cortisol.

MR Protocol: The MR experiments will be performed on the GE 7T whole-body scanner in the Surbeck Laboratory using a 32-channel receive-only array with a 2-channel transmit coil. The MR protocol includes structural images, metabolic imaging, structural and functional connectivities.

ELIGIBILITY:
Inclusion Criteria:

* adolescent participants ages 16-24 yrs old (NIH defines adolescents as up through age 24 years old)
* mild-to-moderate depression with the BDI-II score greater than or equal to 14 (Smarr and Keefer 2011)
* technologically able (Zoom);
* nonpractitioners of daily meditation/breath-work.

Exclusion Criteria:

* pregnant or lactating females
* metal implants unsafe for MRI
* current or lifetime diagnosis of schizophrenia, schizoaffective, bipolar on lithium, or seizure disorders
* recent surgical patient (within 6 months)
* substance use disorder within the last 1 year
* history of significant medical conditions (e.g. traumatic brain injury)
* suicidal ideation (SI) with intent and/or plan to harm self (SI without intent and/or plan to harm self will be allowed to enter the study)

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Depressed adolescents and healthy controls ages 16-24 years old
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Depression Scores on the Beck Depression Inventory-II (BDI-II) | Baseline and 1month, Baseline and 2 months
  The differences at 8-week between intervention and controls in depression and anxiety as measured by the Beck Depression Inventory-II. Twenty-one questions, self reporting with scores ranging from 0 to 63. Higher score indicates more severe depression.
Mean Change in Depression Scores on the Generalized Anxiety Disorder-7. | Baseline and 1month, Baseline and 2 months
  The differences at 8-week between intervention and controls in depression and anxiety as measured by the Generalized Anxiety Disorder-7. Seven questions on a three point scale, a score of 8 or greater represents a reasonable cut-point for identifying probable cases of generalized anxiety disorder.

SECONDARY OUTCOMES:
Mean Change in Reynolds Adolescent Depression Scale (RADS-2) | Baseline and 1month, Baseline and 2 months
  Thirty questions, self-report measures the four basic dimensions of depression: Dysphoric Mood, Anhedonia/Negative Affect, Negative Self-Evaluation, and Somatic Complaints. Identifies depressive symptoms in adolescents, provide an indication of the clinical severity of the individual's depressive symptoms (normal, mild, moderate or severe).
Mean Change in Multidimensional Anxiety Scale for Children (MASC-2) | Baseline and 1month, Baseline and 2 months
  MASC-2 is a self reporting questionnaire with fifty questions that assesses the presence of symptoms related to anxiety disorders in youth. Responses on the MASC 2 are combined to create 11 T-scores: MASC 2 Total Score, Separation Anxiety/Phobias, Generalized Anxiety Disorder (GAD) Index, Social Anxiety (Total, Humiliation/Rejection, Performance Fears), Obsessions & Compulsions, Physical Symptoms (Total, Tense/Restless, Panic), and Harm Avoidance. Higher T-scores indicate more severe and/or a greater number of symptoms.
Mean Change in Hamiliton Anxiety Scale (HAM-A) | Baseline and 1month, Baseline and 2 months
  HAM-A is a fourteen item questionnaire that measure the severity of anxiety symptoms. Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No